CLINICAL TRIAL: NCT00669500
Title: Body Worlds 3 - Nutrition and College of Pharmacy Weeks Exhibit and Lifestyle Intervention
Brief Title: Body Worlds 3 Nutrition Display
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jackilen Shannon, PhD, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: OHSU eIRB3694
Record Dates: First submitted 2008-04-28; First posted 2008-04-30 (Estimated); Last update posted 2011-09-28 (Estimated); Status verified 2011-09

CONDITIONS: Obesity; Hyperlipidemia
Keywords: dietary intake; genetic predisposition; body composition
MeSH Terms: conditions — Obesity; Hyperlipidemias; Genetic Predisposition to Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Lifestyle intervention — Alive!TM web-based, 12 week lifestyle intervention sent via NutritionQuest.

SUMMARY:
Primary Aim # 1: Determine the willingness of the public to participate in an intervention trial - NutritionQuest's Alive!TM - available in a public forum.

Aim #1 Hypotheses: Less than 10% of individuals visiting the NutritionWeek site will register to participate in the Alive!TM Intervention; 70% of these individuals will complete the full intervention.

Primary Aim # 2: To determine among individuals enrolled in the Alive!TM intervention, changes in measurements of body composition from pre- to post-intervention.

Aim #2 Hypotheses: Participation in Alive!TM will result in positive changes in body composition, including reduction of body weight, percent body fat and blood LDL and an increase in blood HDL cholesterol.

Purposes:

1. Educate the public on the relationship between diet, weight and chronic disease
2. Collect data for future research
3. For participants of the Oregon Museum of Science and Industry (OMSI) portion of this study, we also provide a diet assessment and optional 3-month intervention

Recruitment:

Researchers will have a display at OMSI coincidental with the Body Worlds 3 exhibit and at local health fairs. Participants will be recruited from the attendees of the OMSI Body Worlds 3 exhibit as well as general OMSI visitors from July through October 2007 and from health fairs at later dates.

Subject procedures:

No identifiable information will be collected; only gender, year of birth, race and ethnicity are collected on any participant.

Subjects under age 18 can participate in any or all of the following: a brief online, touch-screen assessment of eating and physical activity (health screening for immediate, printed feedback), physiologic measurements (height, weight, hip and waist circumference, percent body fat, blood pressure).

Subjects who are age 18 and over can participate in any or all of the following: a brief online, touch-screen assessment of eating and physical activity (health screening for immediate, printed feedback), physiologic measurements (height, weight, hip and waist circumference, percent body fat, blood pressure), finger prick to assess blood glucose and lipid levels as well as DNA sample (mouthwash swish).

For participants of the OMSI portion of this study, adults may also choose to join a 3-month online lifestyle intervention (Alive!™). Participants who enroll in the 3-month intervention will receive 12 intervention messages over a 3-month period. Each of the messages will take about 5 to 10 minutes to read. At the end of this 3-month period, participants will receive a post-assessment health screening at the Oregon Health & Science University (OHSU) Clinical and Translational Research Center. This post-assessment will include completion of a diet and physical activity assessment, fasting blood measures of glucose and lipids, blood pressure, weight and height.

All visitors to the display area and all research subjects will be offered educational materials.

Instruments used, for OMSI participants only:

The Alive!TM lifestyle intervention is a web-based diet assessment program designed to help individuals evaluate their diet and make healthy changes via tailored e-mail correspondence. This program is operated by NutritionQuest out of Berkeley, California; utilizing the Block questionnaires, designed and validated over many years by Dr. Gladys Block, and now in use by researchers and health practitioners world-wide.

Data analysis:

De-identified data will be stored for future analyses and will be used in descriptive analyses to provide information on the distribution of body size variables and how they relate to reported dietary intake. DNA data from cheek cell samples will be linked by identification number to dietary intake and physiologic measures. Though de-identified, this data may still be used to identify genetic profiles of individuals with various physiologic parameters.

For OMSI participants only:

Alive!TM lifestyle intervention data will be used to determine predictors of change in physiologic and reported intake measures pre and post-intervention, using analysis of variance. At the time of analyses ALL data (including Alive!TM participant data) will be de-identified.

ELIGIBILITY:
Inclusion Criteria:

* Attendees of public health fairs
* General population
* Under the age of 18
* Above the age of 18

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3188 (Actual)
Dates: Start 2007-07; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Determine the willingness of the public to participate in an intervention trial - NutritionQuest's Alive!TM - available in a public forum. | pre-intervention

SECONDARY OUTCOMES:
To determine among individuals enrolled in the Alive!TM intervention, changes in measurements of body composition from pre- to post-intervention. | pre- and post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jackilen Shannon, PhD, Principal Investigator — OHSU Center for Research on Occupational and Environmental Toxicology
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States